CLINICAL TRIAL: NCT04411875
Title: Bioequivalence of Levamlodipine Besylate Tablets in Healthy Chinese Subjects: A Single-dose and Two-period Crossover Study
Brief Title: Bioequivalence of Levamlodipine Besylate Tablets in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 180815-ALDP-01
Record Dates: First submitted 2020-05-19; First posted 2020-06-02 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Healthy Subjects
Keywords: levamlodipine; bioequivalence; pharmacokinetics
MeSH Terms: interventions — Amlodipine; levamlodipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amlodipine (Active Comparator): amlodipine reference formulation at a single dose of 10 mg
  Interventions: Drug: Amlodipine 10 mg
- Levamlodipine (Experimental): levamlodipine test formulation at a single dose of 5 mg
  Interventions: Drug: Levamlodipine 5 mg

INTERVENTIONS:
Drug: Amlodipine 10 mg — The subjects randomly received single oral administration of amlodipine 10 mg.
  Arms: Amlodipine
Drug: Levamlodipine 5 mg — The subjects randomly received single oral administration of levamlodipine 5 mg.
  Arms: Levamlodipine

SUMMARY:
The single-dose randomized, open-label, two-period crossover study was executed in the Phase I Clinical Research Center of the Affiliated Hospital of Qingdao University. According to the random table generate by SAS 9.4, the subjects were divided into two groups at the ratio of 1:1. The select qualified volunteers were hospitalized in the Phase I Clinical Research Center, and fasted for 10 hours overnight until administration. The medicine was swallowed with 240 ml water at room temperature. Blood samples were taken before administration and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 36, 48, 72, 96, 120, 144, 168 hours after administration. The samples were centrifuged at 1,800 g for 10 min at 4 °C to separate the plasma. The plasma samples were divided into two aliquots and stored at -80 °C until bioanalysis. The half-life of levamlodipine is 30 ~ 50 hours. Washout period, the interval between two administration, is 21 days. In the two periods, the operation was kept the same.

Moreover, in high fat meal group, the high-fat breakfast was arranged within half an hour before taking the medicine. Other procedures were the same as those in the fasting group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 18 and above.
* The body mass index is in the range of 18.6-28.5 kg/m2 (including the critical value). The weight of male is not less than 50.0 kg, and that of female is not less than 45.0 kg.
* The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: Vital signs, physical examination, blood routine, blood biochemistry, urinalysis, pregnancy test for female, serological tests for hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), and syphilis virus, 12 lead ECG, breath test for alcohol, drug abuse test.
* The subjects have no family planning within 3 months and could select contraceptive method.
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.

Exclusion Criteria:

* Being allergy to the study medications, smoking, alcohol abuse.
* Participation in another clinical trial within 3 months.

Ages: 19 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 64 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 64 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 64 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 64 days
  Collection of adverse events
Incidence of abnormal blood pressure | 64 days
  Monitor both systolic and diastolic blood pressure
Incidence of abnormal temperature | 64 days
  Monitor the temperature
Incidence of abnormal pulse | 64 days
  Temperature the pulse
Incidence of abnormal electrocardiogram waveform | 64 days
  Electrocardiogram inspection

CONTACTS AND LOCATIONS:
Overall Officials: yu Cao, Doctor, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase Ⅰ Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
The technical achievements (including but not limited to patent right and thesis publishing right) involved in this trial, clinical research materials and achievements are owned by Zhejiang onlycom Pharmaceutical Co., Ltd. With the written consent of Zhejiang onlycom Pharmaceutical Co., Ltd., all partners have the right to publish academic papers, and the Affiliated Hospital of Qingdao University, a clinical research institution, has the right to exchange research results in academic conferences or journals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data have been available on February 15, 2019. The duration has not been determined.

REFERENCES:
- [Derived] Li X, Wang C, Li T, Liu Y, Liu S, Tao Y, Ma Y, Gao X, Cao Y. Bioequivalence of levamlodipine besylate tablets in healthy Chinese subjects: a single-dose and two-period crossover randomized study. BMC Pharmacol Toxicol. 2020 Nov 19;21(1):80. doi: 10.1186/s40360-020-00459-6. PMID 33213527